CLINICAL TRIAL: NCT04603768
Title: Comparison of Theraband, Co-contraction and Isometric Exercises in Patients With Chronic Frozen Shoulder
Brief Title: Comparison of Theraband, Co-contraction and Isometric Exercises in Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1021 Ayesha Zakir
Record Dates: First submitted 2020-10-19; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Frozen Shoulder
Keywords: Theraband; Co-contraction Isometric; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Theraband exercises (Experimental): Group A: baseline physical therapy treatment along with theraband exercises
  Interventions: Other: Theraband exercises
- Co-contraction exercises (Experimental): Group B: baseline physical therapy treatment along with co-contraction exercises
  Interventions: Other: Co-contraction exercises
- isometric exercises (Experimental): Group C: baseline physical therapy treatment along with isometric exercises
  Interventions: Other: Isometric exercises

INTERVENTIONS:
Other: Theraband exercises — Group A performed theraband exercises for 6 weeks.In the first 2 weeks theraband with low resistance was used to perform exercises and then we proceeded gradually with higher resistance therabands.Theraband exercises was performed for Shoulder Flexion,Shoulder Extension Strengthening, Shoulder Internal Rotation Strengthening, Shoulder External Rotation Strengthening, Shoulder Abduction, Empty Can Exercise & Rowing Exercise with 8-10 reps, 3sec hold and 2-3 sets With each of these exercises
  Arms: Theraband exercises
Other: Co-contraction exercises — Muscle co-contraction is the simultaneous contraction of the muscles acting around a joint. Subject stood upright & contracted both the groups (agonist and antagonist) simultaneously without bringing movement at shoulder joint with 6-8 reps , 3sets & 5- 15 seconds duration of sustained self-arm bracing or stiffening was maintained.
  On eligible participants baseline assessment was done,3 session were given 3days per week, post intervention assessment was taken at 3rd and 6th week
  Arms: Co-contraction exercises
Other: Isometric exercises — Isometric exercises of shoulder were performed in subjects for 6 weeks which included isometric Shoulder flexion, shoulder abduction isometric exercise, isometric shoulder external rotation, isometric shoulder internal rotation & isometric shoulder extension with 8-10 reps, 5 sec hold and 2 sets.
  On eligible participants baseline assessment was done,3 session were given 3days per week, post intervention assessment was taken at 3rd and 6th week
  Arms: isometric exercises

SUMMARY:
This project was a Randomized control trial conducted to check the effects of in patients with chronic frozen shoulder theraband, isometric and co-contraction exercises so that we can have best treatment option for patients with chronic frozen shoulder. upper cross syndrome, duration was of 6months,convenient sampling was done, subject following eligibility criteria from DHQ hospital Sheikhupura, were randomly allocated in three groups via lottery method, baseline assessment was done, Group A participants were given baseline treatment along with theraband exercises , Group B participants were given baseline treatment along with co-contraction exercises and Group C were given baseline treatment along with isometric exercises on 3rd and 6th week, post intervention assessment was done via, Numeric pain rating scale(NPRS),Shoulder Pain And Disability Index (SPADI) and goniometric measurements of shoulder ranges ,3 sessions per week were given, data was analyzed by using SPSS version 26.

DETAILED DESCRIPTION:
Frozen shoulder is among the most commonly reported problems to physicians, orthopedics and physical therapists. Even before reporting to clinics there is long history of using over the counter pain killers. Pain avoidance behaviors let the joint stiff so much that a clinician help is sought. Most times the cause of frozen shoulder is not known, therefore is termed as 'idiopathic frozen shoulder'.There is huge literature regarding the management of frozen shoulder and yet after the decades of research there are gaps in treatment options. In modern age of health care, it is common goal of every health care to make patient self-sufficient as early as possible. The self-care models have tremendous advantages. The current study has compared the use of theraband, co-contraction and isometric exercises. The current study was novel in a way that there is limited literature about treating shoulder hypomobility with physical strengthening exercises. All three methods were employed to see if they improve ranges along with accompanying pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic with 6 month chronicity.
* Patients with AROM/PROM less than or equal to 90 degrees.
* Affected shoulder has not more than 90 degrees of abduction & 50% decreased external rotation as compared to normal side/normal ROM values.

Exclusion Criteria:

* Traumatic & diabetic.
* Patient with any cervical or thoracic problem.
* Patients with any intra-articular injection in glenohumeral joint.
* Patients with rotator cuff complete tear.
* Patients with any other serious pathology/red flags

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating scale (NPRS) | 3rd day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain

SECONDARY OUTCOMES:
SPADI | 3rd day
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.

OTHER OUTCOMES:
Goniometric measurement of Shoulder ROM | 3rd day
  A goniometer is an instrument which measures the available range of motion at a joint.Flexion, Extension,Adduction,Abduction, Internal Rotation,External Rotation

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur-Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- DHQ hospital, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan HBY, Pua PY, How CH. Physical therapy in the management of frozen shoulder. Singapore Med J. 2017 Dec;58(12):685-689. doi: 10.11622/smedj.2017107. PMID 29242941
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Moradi M, Hadadnezhad M, Letafatkar A, Khosrokiani Z, Baker JS. Efficacy of throwing exercise with TheraBand in male volleyball players with shoulder internal rotation deficit: a randomized controlled trial. BMC Musculoskelet Disord. 2020 Jun 13;21(1):376. doi: 10.1186/s12891-020-03414-y. PMID 32534582
- [Background] Hanchard N. Exercise classes supervised by a physiotherapist may be better at restoring function after frozen shoulder than individual physiotherapy. J Physiother. 2014 Dec;60(4):236. doi: 10.1016/j.jphys.2014.08.011. Epub 2014 Oct 23. No abstract available. PMID 25439717
- [Background] Lin HC, Li JS, Lo SF, Shih YF, Lo CY, Chen SY. Isokinetic characteristics of shoulder rotators in patients with adhesive capsulitis. J Rehabil Med. 2009 Jun;41(7):563-8. doi: 10.2340/16501977-0378. PMID 19543668
- [Background] Shishir M, Abraham MM, Kanagasabai R, Najimudeen S, Gnanadoss JJ. Home Based Exercise Program for Frozen Shoulder-Follow-up of 36 Idiopathic Frozen Shoulder Patients. Indian Journal of Physiotherapy and Occupational Therapy. 2013;7(3):221.
- [Background] Alptekin HK, Aydin T, Iflazoglu ES, Alkan M. Evaluating the effectiveness of frozen shoulder treatment on the right and left sides. J Phys Ther Sci. 2016 Jan;28(1):207-12. doi: 10.1589/jpts.28.207. Epub 2016 Jan 30. PMID 26957759
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601
- [Background] Sato H, Maruyama H. The Effects of Indirect Treatment of Proprioceptive Neurosmuscular Facilitation. Journal of Physical Therapy Science. 2009;21(2):189-